CLINICAL TRIAL: NCT05820958
Title: The Influence of Intensified Tactile Contact With a Newborn on the Emotional Transformation of Women After Physiological Delivery
Brief Title: Intensified Tactile Contact With a Newborn Andt Emotional Transformation of the Mother
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Jerzy Kukuczka Academy of Physical Education in Katowice (Other)
Responsible Party: Principal Investigator, Rafał Gnat, MSC, associate professor, The Jerzy Kukuczka Academy of Physical Education in Katowice
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 8/2017
Record Dates: First submitted 2023-03-23; First posted 2023-04-20 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Parturition; Depression, Postpartum
Keywords: postpartum; depression; emotional transformation; tactile contact; massage
MeSH Terms: conditions — Depression, Postpartum; Depression

STUDY DESIGN:
Intervention Model Description: In this project, we tested the effect of a single intervention, i.e. intensification of tactile contact between mother and newborn, in the group of volunteers.
  The equivalent control group was selected from participants of our previous, observational study based on a non-random, matched sampling method.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigators were blinded to the results in that way that questionnaires serving as outcome measures were filled up online and results were recorded in the online database. This process was fully automatic. The investigators were unaware of the results until the base was 'opened' after the completion of the study.
  After the completion of the study, the control group was selected from participants of our previous, observational study based on a non-random, matched sampling method. this procedure was completed by one of the investigators. Then, the data were sent to the outcomes assessor with the names of the groups coded. The assessor was unaware of the roles of the two groups in the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The experimental group received an intervention in the form of intensified tactile contact of a mother with the newborn.
  Interventions: Other: Shantali massage
- Control group (No Intervention): The control group received no intervention similar to experimental intervention.

INTERVENTIONS:
Other: Shantali massage — The tactile contact of a mother with the newborn was intensified by means of Shantali massage applied at least 2 times a day, 10 min. Additional, spontaneous sessions were allowed as well. This started on the 3rd day after delivery and lasted until the end of the 12th week after delivery. A total of 169 mandatory sessions should have been provided plus spontaneous sessions, if any.
  The order of application:
  * face and chest; 4 types of movements 10reps each;
  * upper extremity; 4 types of movements, 10 reps each (left and right separately);
  * abdomen; 2 types of movements, 10 reps each;
  * lower extremity; 3 types of movements, 10 reps each (left and right separately);
  * back; 2 types of movements, 10 reps each;
  * final integration; 3 types of movements, 10 reps each.
  Arms: Experimental group

SUMMARY:
The goal of this clinical trial is to test the influence of intensified tactile contact between mother and newborn on the direction of the emotional transformation of the mother from the physiological, undisturbed delivery to 12 weeks postpartum. The participants will deliver intensified tactile stimulation to their newborns in the form of Shantali massage at least 2 times a day. Researchers will compare the results obtained in the intervention group to the control group in which participants voluntarily did not agree to introduce more intensive tactile contact with the child. The main question the study aims to answer is: Is the direction of the mother's emotional transformation different after the intensification of tactile contact with the newborn in comparison to the control group?

DETAILED DESCRIPTION:
Postpartum blues, depression, and psychosis are frequent, burdensome disorders acknowledged by WHO. Investigations into their mechanisms, possible causes, and treatments are strongly needed.

OVERALL RESEARCH QUESTION Is the direction of the mother's emotional transformation different after the intensification of tactile contact with the newborn in comparison to the control group? DESIGN In the study, the non-randomized quasi-experimental design was applied. The dependent variables were: the level of emotions in the designated 'negative' domain (depression, anxiety, negative affects); the level of emotions in the designated 'positive' domain (satisfaction, sense of effectiveness, positive affects). Their values were measured with the use of four standardized, self-reported questionnaires two times, i.e. before and after the 12-week observation period.

PARTICIPANTS The experimental group was selected from the local population of pregnant women who volunteered to provide experimental intervention to their children after birth. Purposive sampling was utilized based on specified eligibility criteria. The intervention (see below) started on the 3rd day after birth and lasted until the end of the 12th week postpartum. Finally, 43 participants completed the procedure.

The control group consisted of the participants from our previous, observational study matched by age, body mass, and height to the participants of the experimental group. These women consciously did not agree to apply the experimental intervention to their children during the observation period.

All participants attended lectures and practical training in a local childbirth school. The volume of their education was similar, except for the training of experimental intervention (5h in total) which was additionally introduced in the participants of the experimental group.

INTERVENTION In the experimental group, the intervention was applied in the form of intensified tactile contact between a mother and the newborn. It was done by means of Shantali massage applied at least in 2 sessions a day, 10 min each. Additional, spontaneous sessions were allowed. This started on the 3rd day after birth and lasted until the end of the 12th week after birth. A total of 169 mandatory sessions should have been provided plus spontaneous sessions, if any. No intervention was applied in the control group.

MEASUREMENTS Four standardized, self-reported psychological questionnaires were used. Their text was digitalized and provided to the participants as an online form. All answers were automatically transported to the digital database. The base was opened after the completion of data collection. Investigators were unaware of the results until that time. They did not have the possibility of exerting any influence on the results during the time of intervention.

PROCEDURE After the recruitment, all participants were thoroughly prepared for delivery in the one childbirth school. They were all supervised by a medical doctor, psychologist, physiotherapist, and nurse at the maternity ward of the one of local hospitals. All procedures were similar in the experimental and control groups (except for normal individualization of the medical/psychological approach). If no postpartum complications occurred, the first measurement of the dependent variables took place on the 3rd day after birth. During the intervention period, participants felt free to contact any member of the specialists mentioned above as well as anyone of the investigators in case of problems, misunderstandings, etc. They started so-called research diaries to record any events that might influence their medical/psychological status during the intervention/observation period (see eligibility criteria). In the experimental group, participants recorded all intervention sessions (both mandatory and spontaneous) they completed. The final measurement of the dependent variables values took place within the 13th week after birth.

STATISTICAL ANALYSIS The internal consistency of the questionnaires was evaluated using the Cronbach alpha coefficient. Inter-group differences were analyzed using the appropriate parametric or non-parametric tests. Cluster analysis was introduced in order to distinguish eventual homogenous subgroups (indicating different directions of postpartum emotional transformation) among participants of both experimental and control groups. Correlations between values of dependent variables were tested as well.

ELIGIBILITY:
Inclusion Criteria:

* first physiological delivery;
* no previous miscarriages;
* normal course of pregnancy;
* normal fetal development confirmed by prenatal ultrasound examination;
* consent to the intervention in the form of intensifying tactile contact with the child during the observation period.

Exclusion Criteria:

* poor health of the child after birth, Apgar score< 8 points;
* complicated physiological delivery with accompanying poor physical condition of the mother after delivery (deep vein thrombosis, pulmonary embolism, postpartum hemorrhage, inflammation);
* deterioration of the child's health condition preventing contact between mother and child (child's illness, incubation of the child);
* deterioration of the mother's health during the observation period;
* deterioration of the mother's emotional state during the observation due to external factors, such as sudden deterioration of the financial situation, traumatic family events (death, severe illnesses, accidents, etc.), significant deterioration of partnership relations between the child's parents, emotionally burdensome legal problems.
* lack of proper compliance with intervention procedures in the form of intensifying tactile contact with the child, the number of procedures performed <50% of the recommended number.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2021-01-10 (Actual); Primary Completion 2022-02-14 (Actual); Study Completion 2022-04-10 (Actual)

PRIMARY OUTCOMES:
Change in Edinburgh Postnatal Depression Scale | 1) 3rd day after delivery; 2) within 13th week after delivery
  Psychological questionnaire used to evaluate the change of postpartum depression level.
  Minimal score - 0 points; maximal score - 30 points. A higher score indicates a higher level of postpartum depression (i.e. higher score = worse).
  The questionnaire was presented to respondents in an online form.
Change in The Hospital Anxiety and Depression Scale | 1) 3rd day after delivery; 2) within 13th week after delivery
  Psychological questionnaire used to evaluate the change in the general level of depression and anxiety associated with the hospital stay.
  Minimal score - 0 points; maximal score - 21 points. A higher score indicates a higher level of depression and anxiety (i.e. higher score = worse).
  The questionnaire was presented to respondents in an online form.
Change in Positive and Negative Affect Schedule questionnaire | 1) 3rd day after delivery; 2) within 13th week after delivery
  Psychological questionnaire used to evaluate the change in the levels of positive and negative affective behavior occurring parallelly in the same person within this same time frame The questionnaire consists of two subscales.
  Subscale 'positive affects':
  Minimal score - 0 points; maximal score - 50 points. A higher score indicates a higher level of positive affects (i.e. higher score = better).
  Subscale 'negative affects':
  Minimal score - 0 points; maximal score - 50 points. A higher score indicates a higher level of negative affects (i.e. higher score = worse).
  The questionnaire was presented to respondents in an online form.
Change in Parenting Sense of Competence questionnaire | 1) 3rd day after delivery; 2) within 13th week after delivery
  Psychological questionnaire used to evaluate the change in the level of parental competence of the respondent The questionnaire consists of two subscales.
  Subscale 'satisfaction':
  Minimal score - 0 points; maximal score - 54 points. A higher score indicates a higher level of parental satisfaction (i.e. higher score = better).
  Subscale 'effectiveness':
  Minimal score - 0 points; maximal score - 48 points. A higher score indicates a higher level of parental effectiveness (i.e. higher score = better).
  The questionnaire was presented to respondents in an online form.

CONTACTS AND LOCATIONS:
Overall Officials: Rafał M Gnat, MSc, Principal Investigator — Rafał Gnat
Locations (1):
- The Jerzy Kukuczka Academy of Physical Education, Katowice, Poland

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD that underlie results in the publication
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 6 months after the publication
Access Criteria: IPD will be shared with the following specialists (based on provided documents confirming their professional status and/or list of publications on the topic or similar topics): physiotherapists, psychologists, psychotherapists, obstetrician MDs, pediatrician MDs.
  Any analyses are allowed provided the original source is clearly indicated in case of any public presentation.
  Requests will be reviewed and answered by the principal investigator.